CLINICAL TRIAL: NCT07302893
Title: Evaluation of an App-Based Sleep Program to Improve Sleep Outcomes in a Clinical Insomnia Population Among New Parents
Brief Title: Evaluation of Digital Sleep Program to Improve Sleep Among New Parents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Udisense DBA Nanit (Industry)
Collaborators: Headspace (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nanit 2025-18
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
Keywords: postpartum; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital CBT-I recipients (Experimental): instructed to follow the 18-session Headspace sleep program daily
  Interventions: Behavioral: Digital CBT-I
- No intervention (No Intervention): asked to maintain their regular routines

INTERVENTIONS:
Behavioral: Digital CBT-I — Headspace 18-session sleep program
  Arms: Digital CBT-I recipients

SUMMARY:
Sleep disturbances are highly prevalent during the postpartum period, with an estimated 40-60% of new parents experiencing inadequate sleep. Although a certain degree of acute sleep disruption is expected after childbirth, excessive or prolonged disturbances can pose significant risks, including poorer cardiometabolic and mental health, impaired cognitive performance, and challenges in bonding with the infant. In addition, untreated insomnia in the perinatal period can lead to more chronic forms of insomnia in some individuals that extends beyond the perinatal period.

Cognitive Behavioral Therapy for Insomnia (CBT-I) is widely recognized as the gold standard treatment for chronic insomnia, demonstrating robust efficacy in diverse populations. However, its applicability in the postpartum period remains underexplored. New parents face a distinct set of sleep challenges, most notably, a significant loss of control over their sleep schedules due to infant care demands. This unpredictability complicates the implementation of core CBT-I techniques such as sleep restriction and stimulus control. Additionally, postpartum parents often experience heightened fatigue, limited time, and cognitive overload, potentially reducing their ability to engage with and retain behavioral or educational interventions.

This study addresses a significant gap in sleep health research by evaluating whether a modified digital CBT-I intervention, enhanced with brief meditation content, can improve self-reported sleep outcomes in new parents. By including both immediate (post-intervention) and longer-term (3-month follow-up) outcomes, the study aligns with broader public health goals of reducing mental health morbidity and improving functioning in the perinatal population.

The Headspace Health Sleep Program is an 18 day program based on CBT-I, which includes the following intervention components: 1) a sleep diary to monitor sleep and associated factors; 2) cognitive interventions to address maladaptive thoughts related to sleep; 3) behavioral interventions to address maladaptive behaviors related to sleep (e.g., sleep hygiene, stimulus control, and sleep restriction); 4) de-arousal techniques (e.g., mindfulness, breathing, and muscle relaxation exercises).

DETAILED DESCRIPTION:
The purpose of the study is to examine the effectiveness of the Headspace Health Sleep Program for improving subjective sleep quality (i.e., self-reported surveys) in a population of new parents with sleep disturbances. The study will employ a 2-arm app-based intervention involving 1 active intervention (i.e., Headspace Health Sleep Program) and a waitlist control for a duration of 3 months.

A set of outcome measures will be used to evaluate the Headspace Health Sleep Program vs. a waitlist control group. The Insomnia Severity Index (ISI) will be used as a primary outcome measure as well as the Sleep Diary. In addition, secondary outcome measures include Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PSS-10) and General Anxiety Disorder-7 (GAD-7). Baseline measures will be taken prior to randomization, and at post-intervention. 3 months following the post-intervention assessment, participants will again be asked to report sleep quality using self-reported surveys.

Eligible participants will complete a one-week baseline assessment period during which they will be provided with a sleep diary. Each morning, they will receive a brief EMA prompt to record sleep-related information from the previous night. Following the 1-week baseline assessment period, participants will be asked to complete baseline questionnaires (i.e., ISI, PSQI, PSS-10, GAD7). They will then be randomized into one of two groups (Headspace Health Sleep Program or waitlist control). Having completed the intervention, participants will be scheduled for the 1-week post-intervention assessment period. Participants will again complete the sleep diary. At the end of this 1-week post-intervention assessment period, participants will complete questionnaires (i.e., ISI, PSQI, PSS-10, GAD7). 3 months following the post-intervention, participants will be asked to complete the sleep diary for a 1-week follow-up assessment period and in addition the ISI, PSQI, PSS-10, and GAD7.

ELIGIBILITY:
Inclusion Criteria:

* First time parents with infants between 4-12 months of age
* Caregiver is over 18 years old
* Caregiver meets clinical threshold for insomnia (11 or greater on the ISI)
* Own a smartphone that can support downloaded apps
* Fluency in English

Exclusion Criteria:

* A diagnosis of any of the following conditions: self-reported schizophrenia, psychosis, depression, self-harm bipolar disorder, seizure disorder, substance use disorder, recent trauma to the head or brain damage, severe cognitive impairment, serious physical health concerns necessitating surgery or with a prognosis of less than 6 months, or pregnancy. Two or more hospitalizations within the past 6 months for psychiatric reasons.
* Prior enrollment in another CBT-I program
* Regular mindfulness meditation practice
* Diagnosed sleep disordered breathing
* Parents of infants with health complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) score | Change from baseline to immediately post-intervention and 3 months follow-up
  The ISI is a measure of sleep disturbance severity. ISI is a 7-item, self-report measure for the evaluation of insomnia. Items in the ISI concern difficulties falling asleep, problems staying asleep, daytime symptoms connected to the sleeping problem, and worrying about sleeping too little. Each item is rated from 0 to 4, giving the rating scale a maximum summed score of 28 points. According to the guidelines for interpretation, 0-7 should be interpreted as no clinically significant insomnia, 8-14 as subthreshold insomnia, 15-21 as clinical insomnia of moderate severity, and 22-28 as severe clinical insomnia.
Sleep Diary | Change from baseline to immediately post-intervention and 3 month follow-up
  Participants will be asked to complete a daily sleep diary for the duration of the 1-week baseline assessment period and the 1-week post-intervention assessment and the 1-week follow-up period. The sleep diary will be used to measure sleep efficiency (SE) and total wake time (TWT). Sleep efficiency will be calculated by dividing the amount of time sleeping in bed by the amount of time spent in bed. Total sleep time will be calculated as the total amount of nightly sleep. In addition, the sleep diary will measure sleep onset latency (SOL), wake after sleep onset (WASO). The sleep diary data will be averaged across one week with a minimum of 4 nights required for inclusion.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to immediately post-intervention and 3 months follow-up
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances. 19 individual items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Higher scores indicate worse sleep quality where poor sleep will be a PSQI total score of > 5.
Perceived Stress Scale (PSS-10) | Change from baseline to immediately post-intervention and 3 months follow-up
  The PSS is a 10-item scale designed to measure the perception of stress within the past month. Participants use a Likert scale with responses ranging from 0 = never to 4 = very often. PSS-10 scores range from 0-40 with higher scores indicating higher perceived stress. Additionally, scores can be categorized as low (0-13), moderate (14-26), and high (27-40) perceived stress.
General Anxiety Disorder-7 (GAD-7) | Change from baseline to immediately post-intervention and 3-months follow-up
  The GAD-7 is a 7-item self-report scale based on the Diagnostic and Statistical Manual of Mental Disorders-IV criteria for generalized anxiety disorder, with items scored from 0 (not at all) to 3 (nearly every day).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanit office, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregated data collected in this project will be de-identified and made available on a shared secured data repository. Results from this project will be shared and disseminated, including manuscripts will be written and submitted for publication in peer-reviewed journals/conferences. All necessary ethical approvals will be obtained.
Time Frame: Data will be made available upon request after dissemination of results.